CLINICAL TRIAL: NCT01674556
Title: Treatment of Pancreatic Adenocarcinoma by Combining Contrast Agent and Gemitabine Under Sonification
Brief Title: Ultrasound-assisted Treatment of Inoperable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/1601
Record Dates: First submitted 2012-07-13; First posted 2012-08-29 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreatic; cancer; adenocarcinoma; Ultrasound; CEUS
MeSH Terms: conditions — Neoplasms; Adenocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast-enhanced ultrasound (CEUS) (Experimental)
  Interventions: Drug: Gemzar

INTERVENTIONS:
Drug: Gemzar — Gemcitabine in combination with ultrasound (US) contrast agent under sonication

SUMMARY:
The investigators primary aim is to increase chemotherapeutic drug uptake in inoperable tumours

The specific sub-objectives of the studies are:

* To quantify tumour sizes and relate it to the patient survival over time, dependent of treatment method.
* To evaluate and compare the toxic effects and safety of gemcitabine in combination with US contrast agent under sonication with gemcitabine alone.
* Develop and validate new ultrasound perfusion algorithms based on burst- replenishment for diagnosis and monitoring of therapy.
* To quantify gemcitabine and its main metabolites in plasma and in circulating mononuclear cells before, during and after pancreatic sonication, and to quantify the concentration of intracellular endogenous nucleotides in circulating mononuclear cells at the same time points.
* To assess plasma and tissue concentrations of gemcitabine, its main metabolites and endogenous nucleotides in those patients where surgical resection can be performed on standard clinical indications.

DETAILED DESCRIPTION:
The primary outcome is monitor for toxicity effect for the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inoperable pancreatic cancer (ICD-10 C25.0-3) at the Department of Surgical Gastroenterology of Haukeland University Hospital, who have volunteered to participate

Exclusion Criteria:

* Patient participated in an investigational study within 30 days prior to study entry (or, if longer, within five half-lives of the last dose of any investigational drug).
* Patient has severe chronic obstructive pulmonary disease or severe chronic asthma.
* Patient has a history of cardiovascular ischemia, acute myocardial infarction or unstable angina within 3 months prior to study entry.
* Patient has a history of any psychiatric disorder or cognitive impairment that would interfere with participation in the study.
* Patient has a known history of Hepatitis B, Hepatitis C or HIV infection.
* Patient requires dialysis or has severely impaired renal function, defined as a serum creatinine > 180 mmol/L at the Screening Visit.
* Patient has severe impairment of liver function, defined as a serum albumin level ≤ 25 g/L and/or a Protrombin Time INR > 2.3 (or APTT > 6 seconds above the upper limit of normal) at the Screening Visit.
* Patient is pregnant or is breast-feeding.
* Patient is allergic to or intolerant of gemcitabine
* Patient is allergic to or intolerant of SonoVue® BRACCO ultrasound contrast agent
* Any reason why, in the opinion of the investigator, the patient should not participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Toxic effects and safety of gemcitabine in combination with US contrast agent under sonication with gemcitabine alone. | Two years
  To evaluate and compare the toxic effects and safety of gemcitabine in combination with US contrast agent under sonication with gemcitabine alone.

SECONDARY OUTCOMES:
tumor size | one year

OTHER OUTCOMES:
tumor size | one year

CONTACTS AND LOCATIONS:
Overall Officials: Georg Dimcevski, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Dimcevski G, Kotopoulis S, Bjanes T, Hoem D, Schjott J, Gjertsen BT, Biermann M, Molven A, Sorbye H, McCormack E, Postema M, Gilja OH. A human clinical trial using ultrasound and microbubbles to enhance gemcitabine treatment of inoperable pancreatic cancer. J Control Release. 2016 Dec 10;243:172-181. doi: 10.1016/j.jconrel.2016.10.007. Epub 2016 Oct 12. PMID 27744037